CLINICAL TRIAL: NCT04871451
Title: An Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of Repeat Intramuscular ABP-450 (prabotulinumtoxinA) Injection for the Treatment of Cervical Dystonia
Brief Title: Extension Study of ABP-19000 to Evaluate Safety and Efficacy of Repeat Treatments of ABP-450 in Cervical Dystonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEON Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABP-19002
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — prabotulinumtoxin A

STUDY DESIGN:
Intervention Model Description: Approximately 60 subjects from ABP-19000 study, irrespective of treatment allocation, will have the option to continue treatment with ABP-450 via intramuscular injection into affected neck muscles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABP-450 - Between Low Dose and High Dose (Experimental): ABP-450 Between Low Dose and High Dose - Intramuscular injections into affected neck muscles with investigator's determined dose within the range of low dose and high dose - 4 injection cycles at 3-month intervals.
  Interventions: Drug: ABP-450

INTERVENTIONS:
Drug: ABP-450 — ABP-450 (prabotulinumtoxinA) contains a 900kDA botulinum toxin type-A complex produced by the bacterium Clostridium botulinum.
  Other Names: prabotulinumtoxinA

SUMMARY:
This Open-label Extension trial will evaluate the safety and efficacy of ABP-450 for the treatment of cervical dystonia in adults. The study will enroll 60 patients across approximately 42 sites in the United States from Phase 2 (ABP-19000) trial. Study subjects who had their initial dose of study drug in the Phase 2 trial, irrespective of treatment allocation, will be eligible to enroll in this OLE study.

DETAILED DESCRIPTION:
This Open-label Extension trial will evaluate the safety and efficacy of ABP-450 for the treatment of cervical dystonia in adults. The study will enroll 60 patients across approximately 42 sites in the United States from Phase 2 (ABP-19000) trial. Study subjects who had their initial dose of study drug in the Phase 2 trial, irrespective of treatment allocation, will be eligible to enroll in this OLE study. Study subjects will receive a predetermined dose of ABP-450 between the Low Dose and High Dose, based on the investigator's discretion and clinical judgment.

ELIGIBILITY:
Inclusion Criteria:

1. Qualified for and had their initial dose of study drug in the ABP-19000 study.
2. Provided written informed consent to being treated for cervical dystonia with ABP-450.
3. Were a male or female patient between 18 and 75 years of age (inclusive) when they entered the ABP-19000 study.
4. Stated willingness to comply with all study procedures, including attendance at the study center for all study visits as scheduled and have technological capabilities to have tele visits.

Exclusion Criteria:

1. Participated in another interventional study during participation in this study.
2. Were a pregnant or lactating female, or female of child-bearing potential not willing to use an acceptable method of contraception (ie, intrauterine device, barrier methods with spermicide, or abstinence).
3. Would not benefit from treatment with ABP-450 for their cervical dystonia, in the investigator's opinion.
4. Viral or other active infection or any medical condition that, in the opinion of the investigator, classifies the patient as unsuitable for participation in the study or patients who do not seem to be in good general health at the time of Day 0 "rollover", and prior to any investigational study drug administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Comella, Principal Investigator — Rush University Medical Center; Joseph Jankovic, Principal Investigator — Baylor St. Luke's Medical Center
Locations (20):
- United States (20):
  - Arizona Neuroscience Research, Phoenix, Arizona
  - Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Neuro Pain Medical Center, Fresno, California
  - Loma Linda University, Loma Linda, California
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - Infinity Clinical Research LLC, Hollywood, Florida
  - Brainstorm Research, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Neurology One, Winter Park, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Michigan State University, East Lansing, Michigan
  - Quest Research Institute - Hunt - PPDS, Farmington Hills, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Cleveland, Ohio
  - The Orthopedic Foundation, New Albany, Ohio
  - Veracity Neuroscience LLC, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data collected during the trial, after deidentification may be shared following review of the clinical study report by the FDA review division and if a decision is made to publish the results in a publication outside posting the results in clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed ABP-19000 study had the option to roll over to this ABP-19002 study at the same site they were previously enrolled.
Pre-assignment Details: Of the 57 who completed ABP-19000 study, 51 participants were dosed and 51were included in the modified full analysis set (mFAS) for the efficacy analysis.
Groups:
- ABP-450 - 150U: ABP-450 Low Dose - Intramuscular injections into affected neck muscles.
- ABP-450 - 250U: ABP-450 Medium Dose - Intramuscular injections into affected neck muscles.
- ABP-450 - 350U: ABP-450 High Dose - Intramuscular injections into affected neck muscles.
Period: Overall Study
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Started | 25 | 17 | 9
Completed | 18 | 15 | 7
Not Completed | 7 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U | Total
Number analyzed (Participants) | 25 | 17 | 9 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (12.72) | 58.0 (10.3) | 52.6 (11.96) | 55.3 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 3 | 34
  Male | 8 | 3 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 0 | 6
  Not Hispanic or Latino | 21 | 15 | 9 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 22 | 16 | 9 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 17 | 9 | 51
Weight (kg) [Mean (Standard Deviation); unit: kg] | 78.71 (15.18) | 73.6 (15.69) | 98.66 (24.84) | 79.86 (18.65)
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.02 (4.69) | 27.22 (4.96) | 31.69 (6.18) | 28.28 (5.13)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Serious Adverse Events
Description: The primary safety endpoint will be the incidence of treatment-related serious adverse events since the start of treatment by Treatment Group when dosed with ABP-450 between Low Dose and High Dose.
Time Frame: Up to 52 weeks
Population: The safety analysis set consisted of all patients who received at least 1 dose of ABP-450. The safety analysis set was used to analyze all safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 25 | 17 | 9
Participants | 0 | 0 | 0

2. Secondary Outcome: Mean Change in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Total Score
Description: The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) scale is used to assess the severity of cervical Dystonia. The TWSTRS-total score has a minimum score of 0 and a maximum score of 85, where higher scores represent worse outcomes. It comprises 3 subscales, which are summated to get the total score: the Torticollis Severity Scale (minimum score of 0, maximum score of 35), the Disability Scale (minimum score of 0, maximum score of 30), and the Pain Scale (minimum score of 0, maximum score of 20).
Time Frame: Four weeks after the dose of each cycle (4 cycles)
Population: Included all patients in the safety analysis set, but excluded patients who had significant changes to their "stable" background medication, received a dose outside the dose range or received alternative or prohibited medications, or did not receive at least 1 treatment of ABP-450 during the OLE study. The number of participants in each treatment cycle could change due to dose multiplication, however for the outcome measure data table the numbers reflect cycle 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 23 | 19 | 4
units on a scale
  Baseline | 41.58 (9.369) | 42.87 (6.631) | 45.63 (5.483)
  Cycle 1, Week 4 | 27.54 (15.873) | 28.47 (12.743) | 34.17 (6.166)
  Cycle 2, Week 4 | 31.17 (15.205) | 24.0 (12.808) | 23.71 (10.917)
  Cycle 3, Week 4 | 28.19 (14.179) | 24.17 (12.302) | 24.82 (9.558)
  Cycle 4, Week 4 | 31.45 (15.666) | 28.6 (11.967) | 27.75 (9.601)

3. Secondary Outcome: Mean Change in the Subscale Score of Severity of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)
Description: The Severity subscale of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) is used to assess the severity of torticollis in cervical dystonia. The severity subscale has a minimum score of 0 and maximum score of 35, where higher scores represent worse outcomes.
Time Frame: Four weeks after the dose of each cycle (4 cycles)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 23 | 19 | 4
units on a scale
  Baseline | 18.8 (3.92) | 19.6 (2.71) | 22.3 (2.22)
  Cycle 1, Week 4 | 12.6 (6.38) | 14.0 (4.97) | 19.3 (1.53)
  Cycle 2, Week 4 | 15.3 (5.56) | 11.0 (6.55) | 14.4 (5.71)
  Cycle 3, Week 4 | 12.1 (5.59) | 11.1 (6.44) | 13.6 (5.97)
  Cycle 4, Week 4 | 12.6 (6.39) | 14.8 (4.96) | 15.8 (5.64)

4. Secondary Outcome: Mean Change in the Subscale Score of Disability of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Spasmodic Torticollis Rating Scale (TWSTRS)
Description: The Disability subscale of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) is used to assess the severity of disability in cervical dystonia. The disability subscale has a minimum score of 0 and maximum score of 30, where higher scores represent worse outcomes.
Time Frame: Four weeks after the dose of each cycle (4 cycles)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 23 | 19 | 4
units on a scale
  Baseline | 11.2 (4.78) | 11.9 (4.17) | 12.5 (2.89)
  Cycle 1, Week 4 | 6.9 (6.75) | 7.8 (5.29) | 9.0 (2.65)
  Cycle 2, Week 4 | 8.8 (6.68) | 6.7 (5.43) | 5.0 (4.12)
  Cycle 3, Week 4 | 9.1 (5.62) | 6.7 (4.58) | 5.4 (2.94)
  Cycle 4, Week 4 | 9.6 (5.81) | 6.8 (5.71) | 6.2 (5.42)

5. Secondary Outcome: Mean Change in the Subscale Score of Pain of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)
Description: The Pain subscale of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) is used to assess the severity of pain in cervical dystonia. The pain subscale has a minimum score of 0 and maximum score of 20, where higher scores represent worse outcomes.
Time Frame: Four weeks after the dose of each cycle (4 cycles)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 23 | 19 | 4
units on a scale
  Baseline | 11.576 (3.0697) | 11.342 (3.0824) | 10.875 (2.7195)
  Cycle 1, Week 4 | 8.060 (5.1386) | 6.639 (5.1071) | 5.833 (4.7719)
  Cycle 2, Week 4 | 7.167 (5.3940) | 6.333 (3.8441) | 4.286 (2.9595)
  Cycle 3, Week 4 | 6.938 (4.6209) | 6.348 (4.4573) | 5.821 (4.3702)
  Cycle 4, Week 4 | 9.250 (4.5104) | 6.904 (3.9112) | 5.750 (2.7884)

6. Secondary Outcome: Mean Change in Patient Global Impression of Change (PGI-C)
Description: The Patient Global Impression of Change (PGI-C) enables the patient to rate changes in their perception of their general health status over the duration of the assessment via a 7-point scale ranging from "much improved" to "much worse". The 7-point scale range is much improved (+3) to much worse (-3) with no change at "0". For the analysis, the data was transformed to a linear 7 point scale where 1 = much better and 7 = much worse.
  The mean change in the subject's assessment of the change in clinical status since the start of treatment measured by the Patients' Global Impression of Change (PGI-C) Scale was assessed by Treatment Group at Week 4.
Time Frame: Four weeks after the dose of each cycle (4 cycles)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 23 | 19 | 4
units on a scale
  Baseline | 3.8 (1.68) | 4.1 (1.35) | 3.8 (2.36)
  Cycle 1, Week 4 | 2.1 (1.14) | 2.2 (1.17) | 1.7 (0.58)
  Cycle 2, Week 4 | 2.2 (1.53) | 2.4 (1.63) | 1.6 (0.79)
  Cycle 3, Week 4 | 1.8 (0.89) | 2.4 (1.47) | 1.9 (0.69)
  Cycle 4, Week 4 | 1.8 (0.84) | 1.4 (0.77) | 2.0 (0.63)

7. Secondary Outcome: Mean Change in Clinical Global Impression of Change (CGI-C)
Description: The Clinical Global Impression of Change (CGI-C) enables the patient to rate changes in their perception of their general health status over the duration of the assessment via a 7-point scale ranging from "much improved" to "much worse". The 7-point scale range is much improved (+3) to much worse (-3) with no change at "0". For the analysis, the data was transformed to a linear 7 point scale where 1 = much better and 7 = much worse.
  The mean change from Baseline in the Clinical Global Impression of Change (CGI-C) Score was assessed by Treatment Group at Week 4.
Time Frame: Four weeks after the dose of each cycle (4 cycles)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 23 | 19 | 4
units on a scale
  Baseline | 3.4 (1.44) | 3.7 (1.37) | 3.8 (1.71)
  Cycle 1, Week 4 | 2.1 (0.94) | 1.9 (0.94) | 1.7 (0.58)
  Cycle 2, Week 4 | 2.5 (1.24) | 2.0 (1.52) | 1.7 (0.76)
  Cycle 3, Week 4 | 2.1 (0.83) | 2.2 (1.15) | 1.9 (0.69)
  Cycle 4, Week 4 | 2.0 (0.71) | 1.8 (0.60) | 1.8 (0.75)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Arm/Group | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/17 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/17 | 0/9
Other Adverse Events (participants affected / at risk) | 16/25 | 15/17 | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABP-450 - 150U (N=25) | ABP-450 - 250U (N=17) | ABP-450 - 350U (N=9)
COVID-19 (Infections and infestations) | 6 | 4 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 0
Upper Respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 1 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Paresthesia (Nervous system disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood Cholesterol Increased (Investigations) | 0 | 2 | 1
Injection site pain (General disorders) | 3 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT04871451/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT04871451/SAP_001.pdf